CLINICAL TRIAL: NCT06912958
Title: Efficacy of Matcha Tea on Patients With Biofilm-induced Gingivitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Talib (Other)
Responsible Party: Sponsor-Investigator, Ahmed Talib, Clinical researcher, University of Baghdad
Organization: University of Baghdad (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Matcha tea on gingivitis
Record Dates: First submitted 2025-03-27; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Intervention Model Description: The first group recieve the drug A. While the second group will recieve drug B
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Matcha tea group (Experimental): Intake of two cups daily for a month of matcha tea with oral hygiene instructions.
  Interventions: Dietary Supplement: Drinking of matcha tea; Dietary Supplement: Organic Japanese Matcha, Jade Leaf, Japan
- Control group (No Intervention): Oral hygiene instructions, which include brushing teeth and flossing twice daily.

INTERVENTIONS:
Dietary Supplement: Drinking of matcha tea — Japanese tea that will take twice daily for one month
  Arms: Matcha tea group
Dietary Supplement: Organic Japanese Matcha, Jade Leaf, Japan — dietary intake
  Other Names: Lot T47I10P100
  Arms: Matcha tea group

SUMMARY:
1. Evaluate the salivary level of antioxidants (malondialdehyde "MDA," superoxide dismutase "SOD," and glutathione peroxidase-1 "GPX-1") by enzyme-linked immunosorbent assay test (ELISA).
2. Measuring clinical periodontal parameters, which are plaque index (PI), bleeding on probing (BOP), and gingival index (GI), between the baseline and endpoint of the study, which is one month.

DETAILED DESCRIPTION:
Gingivitis is the most common form of periodontal disease (PD). In a survey conducted in three Latin American cities, gingivitis was detected in approximately 99.6% of 1650 subjects. It is defined as inflammation affecting gingival tissue surrounding teeth. Clinically, it is characterized by gingival redness and edema with no periodontal attachment loss.

The generation of reactive oxygen species (ROS) and other free radicals (R) during metabolism is a normal process that ideally is compensated by an endogenous antioxidant system. However, due to many environmental, lifestyle, and pathological situations, excess radicals can accumulate, resulting in oxidative stress. Oxidative stress (OS) has been related to cardiovascular disease, cancer, and other chronic diseases. It also plays an important role in the pathogenesis of periodontal disease.

Inflammatory response is a part of many diseases. It may lead to the production of excessive amounts of substances promoting the production of reactive oxygen species (ROS), which can damage cell structures and lead to long-term disruption in the functioning of the body.

One solution to keeping the appropriate oxidative balance is a high supply of exogenic antioxidants that aims to equalize and prevent oxidative processes. It is also important to maintain a correct lifestyle, free from stress-inducing factors.

There are 3 main varieties of tea: green, black, and oolong. The difference is in how the teas are processed. Green tea is made from unfermented leaves and reportedly contains the highest concentration of powerful antioxidants called polyphenols.

Antioxidants are substances that fight free radicals, damaging compounds in the body that change cells, damage DNA, and even cause cell death. Antioxidants, such as polyphenols in green tea, can neutralize free radicals and may reduce or even help prevent some of the damage.

Matcha tea is Japanese powdered green tea that is derived from the Camellia sinensis plant, the same plant of green tea. It contains huge amounts of polyphenols, amino acids (mainly tannins), and caffeine that probably increase its antioxidant characteristic.

Matcha tea is planted and processed differently. First, during the cultivation, green tea is grown in the sun; however, matcha tea is grown under shadow during the last few weeks before harvesting. Therefore, this difference in cultivation procedure leads to a higher amount of theanine and polyphenols in the content of Matcha tea.

Matcha tea contains more than double the amount of vitamin C than green tea. Vitamin C is a powerful exogenous antioxidant that reinforces the immune defense of the body. Additionally, it helps to seal blood vessels, has anti-inflammatory properties, and also supports the immune system.

ELIGIBILITY:
Inclusion Criteria:

* Having at least 20 teeth.
* gingivitis patient ( BOP<10% , PPD = or <3mm , no CAL , Have plaque index =1 ( according to Quigley-hein plaque index )
* No history of systemic disease.
* No medical treatment that impact periodontal status at last 6 months before examination and sampling.
* life style control

Exclusion Criteria:

* *pregnant or in the period of breast feeding.

  * smokers and alcoholics.
  * Patients wearing orthodontic appliances.
  * has history of systemic disease.
  * periodontitis patient

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-11-17 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-02-04 (Actual)

PRIMARY OUTCOMES:
Evaluate the antioxidant effects of Matcha tea in daily intake for gingivitis patients. | One month
  Evaluate the salivary level of antioxidants (malondialdehyde "MDA," superoxide dismutase "SOD," and glutathione peroxidase-1 "GPX-1") by enzyme-linked immunosorbent assay test (ELISA).

SECONDARY OUTCOMES:
Measuring the changes in the clinical periodontal parameters | one month
  Measuring clinical periodontal parameters, which are plaque index (PI), bleeding on probing (BOP), and gingival index (GI), between the baseline and endpoint of the study, which is one month.

CONTACTS AND LOCATIONS:
Locations (1):
- Baghdad university, Baghdad, City of Medicine, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] (Carr A.C et al ,2017)
- [Background] (Jakubczyk K et al ,2020)
- [Background] (Lobo et al, 2010